CLINICAL TRIAL: NCT01501097
Title: A Randomized Controlled Trial on the Impact of Early Application of CRRT on the Outcomes of Burn Patients With Early Phase of Sepsis
Brief Title: The Impact of Continuous Renal Replacement Therapy on the Outcomes of Burn Patients With Early Phase of Sepsis
Acronym: CRRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Zhiqiang Yuan, Associate Professor, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWHCBS01
Record Dates: First submitted 2011-12-20; First posted 2011-12-29 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Burns; Sepsis
MeSH Terms: conditions — Burns; Sepsis | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention)
  Interventions: Procedure: Continuous Renal Replacement Therapy
- early HV-crrt (Experimental)
  Interventions: Procedure: Continuous Renal Replacement Therapy

INTERVENTIONS:
Procedure: Continuous Renal Replacement Therapy — Patients will be randomized to either arm :early HV-crrt(50ml/kg/h) or Control group

SUMMARY:
The purpose of this study is to determine if early application of CRRT will result in an improvement of clinical outcomes of burn patients during the early phase of sepsis

DETAILED DESCRIPTION:
The impact of Continuous Renal Replacement Therapy (CRRT) on the outcomes of patients with sepsis is controversial, and there is no consensus for the timing and dose of CRRT may improve the outcomes. The purpose of this prospective randomized study is to assess the effect of different CRRT intensity (25ml/kg/h or 50ml/kg/h) on the outcomes of burn patients with early phase of sepsis

ELIGIBILITY:
Inclusion Criteria:

* patients with documented sepsis
* clinically identified focus of infection associated with at least 2 SIRS -criteria and one or more sepsis-induced organ failures within the 24 hours -prior to inclusion
* age 18 to 70 years
* severe burned patients with 50% < TBSA < 85%

Exclusion Criteria:

* cirrhosis child class C
* too high APACHE II & SOFA score at admission
* age over 70 years
* were presence of a malignant tumor, chronic renal insufficiency (serum creatinine > 133 µmol/L), moribund state, receiving immunosuppressive therapy or receiving any kind of renal replacement therapy before randomization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Changes in serum cytokine concentrations and clearance | 96 hours
  0, 6, 12 , 24, 48, 96 hours post CRRT

SECONDARY OUTCOMES:
28 and 90 days survival | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China